CLINICAL TRIAL: NCT04635852
Title: Effentora® for Dyspnoea - Fentanyl Buccal Tablet for the Relief of Episodic Breathlessness in Cancer Patients: A Multicenter, Open Label, Randomized, Morphine-controlled, Crossover, Phase II-TRIAL
Brief Title: Fentanyl Buccal Tablet for the Relief of Episodic Breathlessness in Cancer Patients
Acronym: EFFENDYS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Steffen Simon, prof, University of Cologne
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln-1412; 2011-005797-32 (EudraCT Number); DRKS00004353 (Other: DRKS)
Record Dates: First submitted 2014-01-10; First posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Cancer; Dyspnea, Paroxysmal
MeSH Terms: conditions — Neoplasms; Dyspnea, Paroxysmal | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental): Fentanyl buccal tablet Dosage: 100µg - 600 µg Fentanyl (to be determined by titration) Administration: buccal administration (tablet)
  Interventions: Drug: Fentanyl
- Immediate release morphine (Active Comparator): Immediate release morphine, solution Dosage: Start with a minimum of 5mg (to be determined by titration)
  Interventions: Drug: Immediate release morphine

INTERVENTIONS:
Drug: Fentanyl
  Other Names: Fentanyl buccal tablet; Fentanyl citrate
  Arms: Fentanyl
Drug: Immediate release morphine
  Other Names: Morphine Solution
  Arms: Immediate release morphine

SUMMARY:
"Episodic breathlessness (or dyspnea) is one form of chronic refractory breathlessness characterized by a severe worsening of breathlessness intensity or unpleasantness beyond usual fluctuations in the patient's perception. Episodes are time-limited (seconds to hours) and occur intermittently, with or without underlying continuous breathlessness. Episodes may be predictable or unpredictable, depending on whether any trigger(s) can be identified. There is a range of known triggers which can interact (e.g. exertion, emotions, comorbidities or external environment). One episode can be caused by one or more triggers." ( definition by an international expert consensus [Simon et al. 2013]). Approximately half of patients with cancer complain about breathlessness with the highest prevalence in pulmonary malignancies. Episodic breathlessness is reported by 81% of breathless cancer patients with significant impairment on quality of life and limitations on activity. Although episodic breathlessness show some similar characteristics like episodes of pain (breakthrough cancer pain, BTCP; median duration 30minutes), they are often shorter: 91% last less than 20minutes (min). Other evidence supports these findings with duration between 2-15minutes which is a real challenge for the treatment of episodic breathlessness. In the majority of cases, episodic breathlessness occur 1-4 times per day and peak intensity is rated moderate or severe.

There is evidence for the effectiveness of opioids for the relief of chronic refractory breathlessness. There is no evaluated and proven standard treatment for the relief of episodic breathlessness at the moment but immediate-release morphine (IRM) as solution or tablet is most frequently used in clinical practice to treat episodic breathlessness. Time to onset of action of IRM is about 20-30min for pain. Fentanyl is a potent opioid and shows good evidence for the treatment of BTCP through its quick onset of action (5-15min) and short duration of action (50-60min). Because of its pharmacodynamic properties fentanyl might be appropriate and effective for the relief of episodic breathlessness. However, the efficacy of fentanyl for the relief of breathlessness and time to onset is unknown.

This pilot study aims to evaluate relative efficacy, feasibility and time to onset of two different opioids (fentanyl and morphine) in order to improve the management of episodic breathlessness.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically proven cancer of any entity which is non-curable as judged by the referring physician or investigator
2. To be an inpatient during the study
3. Refractory breathlessness - this study applies only to 'refractory breathlessness ' and is defined: a patient is still breathless although the underlying disease (e.g. lung cancer) or cause of breathlessness (e.g. pleural effusion) is treated optimal as judged by the referring physician or investigator
4. History of recurrent episodic breathlessness - episodic breathlessness is defined as an increase in breathlessness occurring intermittently in patients with or without underlying continuous breathlessness
5. Peak intensity of episodic breathlessness ≥ 3 (NRS, 0-10)
6. Opioid tolerance for at least one day - opioid tolerance is defined: patient who receive per day at least 30mg oral morphine, 15mg oral oxycodone, 4mg oral hydromorphone, 12µg/h transdermal fentanyl or an analgetic equivalent of a different opioid or a different routes of application
7. Life expectancy of at least one month as judged by the referring physician or investigator

Exclusion criteria:

1. Uncontrolled breathlessness (i.e. rapidly worsening breathlessness requiring urgent medical or technical intervention)
2. Uncontrolled performance status (i.e. rapid deterioration of performance status)
3. Consideration of any reason by the referring therapeutic team that the patient is not an appropriate participant of a clinical trial
4. Respiratory depression or preconditions with risk of respiratory depression
5. Acute abdomen or ileus or any situation that drug resorption is not possible
6. Renal dysfunction with creatinine clearance (eGFR) calculated as less than 25 ml/minute
7. Medical history of severe hepatic impairment
8. The use of fentanyl transmucosal products for breakthrough cancer pain (BTCP) during the trial
9. The use of a monoamine oxidase inhibitors within the previous 14 days
10. Treatment with any other investigational drugs within the previous 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to onset of meaningful breathlessness relief | minutes (by stop watch) from drug application of FBT/IRM up to breathlessness relief
  To determine the time to onset of meaningful breathlessness relief of fentanyl buccal tablet (FBT) in comparison to immediate-release morphine (IRM)

SECONDARY OUTCOMES:
Breathlessness intensity | at 0, 3, 5, 10, 15, 20, 30, 45 and 60 minutes after application of FBT/IRM
  Breathlessness intensity measured by NRS (range 0-10)
Numbers of rescue medication doses | Numbers of rescue medication doses through study completion, assessed at day 10 (final visit)
  If adequate breathlessness relief was not reached after 30 min, the patient could use his standard rescue medication.
Patient's & investigator's satisfaction | through study completion, day 10 (e.g. final visit)
  Patient's and investigator's satisfaction of breathlessness relief and route of application regarding ease of administration (4-point verbal rating scale: 0 = poor/unsatisfied and 4 = excellent/very satisfied).
Preferences of study drugs | through study completion, day 10 (e.g. final visit)
  FBT or IRM or both/none

OTHER OUTCOMES:
Number of (serious) adverse events (AE/SAE; Safety of FBNT/IRM) | through study completion, day 10 (e.g. final visit)
  Counts of adverse events
Severity of AE/SAE (Safety of FBNT/IRM) | through study completion, day 10 (e.g. final visit)
  CTCAE tool v4.03 (National Cancer Institute Common Terminology Criteria)
Oxygen saturation (Safety of FBNT/IRM) | through study completion, day 10 (e.g. final visit)
  finger clip pulse oximetry (Contec Medical Systems Co., China)
Patient's vigilance (Safety of FBNT/IRM) | through study completion, day 10 (e.g. final visit)
  Glasgow Coma Scale (GCS)
Respiratory rate (Safety of FBNT/IRM) | through study completion, day 10 (e.g. final visit)
  breaths per minute
Enrollment rate (Feasibility of study procedures) | day 10 (e.g. final visit)
  Ratio of patients screened to patient with informed consent
Completion rate (Feasibility of study procedure) | day 10 (e.g. final visit)
  Ratio of patients that were randomly assigned to the experimental vs active comparator arm to patients that completed the study
Drop outs (Feasibility of study procedures) | day 10 (e.g. final visit)
  Counts of drop out per visit (TPh+EPh)
Reasons for rejection of study participation of screened patient (Feasibility of study procedures) | day 10 (e.g. final visit)
  List of reasons/ free text responses
Acceptability of study procedures | day 10 (e.g. final visit)
  closed questions: 4-point verbal rating scale between 0=poor/unsatisfied and 4=excellent/very satisfied, and yes/no; reports by patients, investigators and clinical team
Acceptability of measurement tools | day 10 (e.g. final visit)
  closed questions: 4-point verbal rating scale between 0=poor/unsatisfied and 4=excellent/very satisfied, and yes/no; reports by patients, investigators and clinical team
Acceptability of rescue procedures | day 10 (e.g. final visit)
  closed questions: 4-point verbal rating scale between 0=poor/unsatisfied and 4=excellent/very satisfied, and yes/no; reports by patients, investigators and clinical team

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Voltz, Professor, Principal Investigator — Department of Palliative Medicine
Locations (3):
- Germany (3):
  - University Hospital Göttingen Center of Palliative Medicine, Göttingen, Hesse
  - Study Center Palliative Medicine, Cologne, North Rhine-Westphalia
  - Hospital Essen- Mitte, Departement of Palliative Medicine, Essen, North Rhine-Westphalia